CLINICAL TRIAL: NCT05997628
Title: The Exploratory Study on the Baseline Level of NAD+/NADH in Peripheral Blood Samples of Different Gender and Age Groups of Healthy Adults.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Collaborators: Shanghai Mengchao Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CH2301-A-01
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: NAD+/NADH in Peripheral Blood Monitoring
Keywords: NADH; NAD+

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18-40 years: Each group has 20 subjects, and the sex ratio of 18-40 years group is 1:1. After each participant is enrolled, peripheral blood samples are taken before breakfast and before lunch to detect NAD+/NADH levels in peripheral blood and determine the physiological baseline levels of NAD+/NADH in different age groups
  Interventions: Other: Detection of NAD+/NADH concentration of Peripheral Blood Samples
- 41-60 years: Each group has 20 subjects, and the sex ratio of 41-60 years group is 1:1. After each participant is enrolled, peripheral blood samples are taken before breakfast and before lunch to detect NAD+/NADH levels in peripheral blood and determine the physiological baseline levels of NAD+/NADH in different age groups
  Interventions: Other: Detection of NAD+/NADH concentration of Peripheral Blood Samples
- 61-80 years: Each group has 20 subjects, and the sex ratio of 61-80 years group is 1:1. After each participant is enrolled, peripheral blood samples are taken before breakfast and before lunch to detect NAD+/NADH levels in peripheral blood and determine the physiological baseline levels of NAD+/NADH in different age groups
  Interventions: Other: Detection of NAD+/NADH concentration of Peripheral Blood Samples

INTERVENTIONS:
Other: Detection of NAD+/NADH concentration of Peripheral Blood Samples — Peripheral blood samples are taken before breakfast and before lunch to detect NAD+/NADH levels, hematology, blood biochemical indicators, immune cells and SIRT1 level in peripheral blood in different age groups. This experiment monitors indicators mentioned above without any drug intervention.

SUMMARY:
This study investigates the concentration levels of NAD+/NADH in peripheral blood samples and immune cells of healthy adults of different age groups under daily physiological and lifestyle conditions, in order to determine the baseline levels of NAD+/NADH in adult populations of different age groups and genders. Simultaneously examining the biological status and function of human immune cells, blood biochemistry, biological age levels, to explore the biological function and mechanism of NAD+/NADH in the aging process of the human body.

DETAILED DESCRIPTION:
In this study, 60 subjects will be enrolled in three groups according to the age range of 20-40, 41-60 and 61-80. Each group has 20 subjects, and the sex ratio of each group is 1:1. After each participant is enrolled, peripheral blood samples are taken before breakfast and before lunch to detect NAD+/NADH levels in peripheral blood and determine the physiological baseline levels of NAD+/NADH in different age groups. At the same time, the subjects tested Hematology, blood biochemical indicators, as well as the expression of subsets of peripheral blood immune cells and SIRT1 level at the same time point, to study the change trend of NAD+/NADH level in different age groups, and the correlation between this trend and Hematology age, immune indicators.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male/females of 18 to 85 years of age.

  2. Able to provide written Informed Consent.

  3. Body Mass Index ranging from 18 to 25 kg/m2(bounds included), with a stable weight over the last 2 months (±2.5 kg).

  4. Able to follow verbal and written study directions.

  5. Must not be taking or be willing to take any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.

  6.Able to maintain consistent diet and lifestyle habits according to the study

Exclusion Criteria:

* 1. Male/females of 18 to 85 years of age.

  2. Able to provide written Informed Consent.

  3. Body Mass Index ranging from 18 to 25 kg/m2(bounds included), with a stable weight over the last 2 months (±2.5 kg).

  4. Able to follow verbal and written study directions.

  5. Must not be taking or be willing to take any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.

  6. Able to maintain consistent diet and lifestyle habits according to the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults of different age groups under daily physiological and lifestyle conditions
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The baseline in NAD+ and NADH concentrations in whole blood of healthy adults. | Fasting at 0 hour, 4 hour on the day of the trial
  Monitor
Counting of blood cell indicators such as red blood cells, white blood cells, and platelets in healthy adults | Fasting at 0 hour on the day of the trial
  Monitor
Blood biochemical indicators of the healthy adults monitoring including liver function; lood lipids; blood sugar; renal function; uric acid; lactate dehydrogenase; creatine kinase, etc | Fasting at 0 hour on the day of the trial
  Monitor
Peripheral blood immune cell phenotype of the healthy adults monitoring including NK cells, B lymphocytes, eosinophils, T lymphocytes, platelet neutrophils, basophils, and monocytes, etc | Fasting at 0 hour on the day of the trial
  Monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR